CLINICAL TRIAL: NCT03140644
Title: SARCOLOWDOSE : Ultra-low Dose CT Scan and MRI in Thoracic Sarcoidosis
Acronym: SARCOLOWDOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-A01781-50; 35RC16_9760 (Other: CHU Rennes)
Record Dates: First submitted 2017-04-25; First posted 2017-05-04 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Sarcoidosis, Pulmonary
Keywords: thoracic sarcoidosis; ultra-low dose computed tomography; Magnetic resonance imaging using Ultrashort echo time
MeSH Terms: conditions — Sarcoidosis, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with thoracic sarcoidosis (Experimental): Patients routinely followed-up for thoracic sarcoidosis with a CT scan indicated in the follow-up
  Interventions: Other: Patients with thoracic sarcoidosis

INTERVENTIONS:
Other: Patients with thoracic sarcoidosis — Ultra-low dose CT scan and MRI with UTE

SUMMARY:
The goal of this study is to evaluate the diagnostic agreement between, on the one hand, ultra-low dose CT and MRI with UTE pulse sequences, and on the other hand, standard CT scan, to quantify lung parenchyma patterns in thoracic sarcoidosis.

DETAILED DESCRIPTION:
Sarcoidosis is a chronic disease involving lung and mediastinum in more than 90% of cases. Five to 25% of thoracic sarcoidosis are complicated by a severe fibrotic lung disease. Computed tomography (CT) is critical for the diagnosis of thoracic sarcoidosis as well as for therapeutic management. Repeated CT examinations, sometimes all life long, raise the issue of the cumulative radiation dose and subsequent risk of cancer, thus pushing the need for imaging techniques using low or no radiation dose. Based upon tube voltage and current reduction as well as iterative recontsruction, ultra-low dose CT (ULD CT) allows to lower the dose up to that of a traditional chest X-ray. Magnetic resonance imaging (MRI) using Ultrashort echo time (UTE) enables lung parenchyma imaging with high signal-to-noise and spatial resolution.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or more
* Diagnosed with thoracic sarcoidosis according to ATS/ERS/WASOG 1999 criteria, with stages 2, 3 or 4, or lung function significantly impaired
* For whom a chest CT examination without contrast medium is indicated in the normal follow-up of the disease
* covered by social security
* having received information about the study and having given written informed consent

Exclusion Criteria:

* Pregnant woman
* Adult person unable to give consent
* Patient in exclusion period du to another protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Percentage of fibrosis within the 2 lungs (reticulations with or without honeycombing) in standard CT and ULD CT to study diagnostic agreement between these techniques | Day 0

SECONDARY OUTCOMES:
Percentage of ground-glass opacity within the 2 lungs in standard CT and ULD CT | Day 0
Percentage of consolidation within the 2 lungs in standard CT and ULD CT | Day 0
Percentage of pulmonary nodules within the 2 lungs in standard CT and ULD CT | Day 0
Percentage of fibrosis within the 2 lungs in standard CT and UTE MRI | Day 0
Percentage of ground-glass opacity within the 2 lungs in standard CT and UTE MRI | Day 0
Percentage of consolidation within the 2 lungs in standard CT and UTE MRI | Day 0
Percentage of pulmonary nodules within the 2 lungs in standard CT and UTE MRI | Day 0
Main pulmonary artery to ascending aorta diameter ratio measured with standard CT | Day 0
Main pulmonary artery to ascending aorta diameter ratio measured with ULD CT | Day 0
Main pulmonary artery to ascending aorta diameter ratio measured with UTE MRI | Day 0
Drent score adapted from Oberstein with standard CT | Day 0
Drent score adapted from Oberstein with ULD CT | Day 0
Drent score adapted from Oberstein with UTE MRI | Day 0
Percentage of fibrosis measured by 2 readers for standard CT | Day 0
Percentage of fibrosis measured by 2 readers for ULD CT | Day 0
Percentage of fibrosis measured by 2 readers for UTE MRI | Day 0
Image quality of lung parenchyma assessed quantitatively using standard CT | Day 0
  signal-to-noise and contrast-to-noise ratios
Image quality of lung parenchyma assessed quantitatively using ULD CT | Day 0
  signal-to-noise and contrast-to-noise ratios
Image quality of lung parenchyma assessed quantitatively using UTE MRI | Day 0
  signal-to-noise and contrast-to-noise ratios
Image quality of lung parenchyma assessed qualitatively using standard CT | Day 0
  4-level scale
Image quality of lung parenchyma assessed qualitatively using ULD CT | Day 0
  4-level scale
Image quality of lung parenchyma assessed qualitatively using UTE MRI | Day 0
  4-level scale
Score of tolerance for CT examinations | Day 0
Score of tolerance for MRI examinations | Day 0

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CH de Bobigny, Hôpital Avicenne, Bobigny
  - CHU de Brest, Brest
  - CH de Lorient, Lorient
  - CHU de Nantes, Nantes
  - CHU Rennes, Rennes
  - CH de Saint-Brieuc, Saint-Brieuc
  - CH de Vannes, Vannes

IPD SHARING:
Plan to Share IPD: No